CLINICAL TRIAL: NCT02074332
Title: Development and Application of Appropriate Technology for Obesity Prevention and Control -- Study on Personalized Aerobic and Appropriate Exercise Technology
Brief Title: Study on Obesity Intervention With Physical Exercise Among Students in Changping District, Beijing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hai-Jun Wang (Other)
Responsible Party: Sponsor-Investigator, Hai-Jun Wang, Professor, Peking University
Organization: Peking University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00001052-12046
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Pediatric Obesity
Keywords: Obesity; Physical activity; Schoolchildren; Intervention Studies
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Intervention (Experimental): Physical activity guidance Health education
  Interventions: Behavioral: Physical activity guidance; Behavioral: Health education
- Control (No Intervention): Receive no intervention

INTERVENTIONS:
Behavioral: Physical activity guidance — Physical education class amelioration Additional physical activities for overweight&obese students Family physical activities Parent involvement
  Other Names: Physical activity programme
  Arms: Intervention
Behavioral: Health education — Knowledge of obesity prevention and control
  Arms: Intervention

SUMMARY:
The primary objective of this study is to assess the effectiveness of a school based physical activity programme on obesity and related health outcomes in young schoolchildren.

ELIGIBILITY:
Inclusion Criteria:

* Grade of 2 to 5 in elementary schools and grade of 1 to 2 in middle schools.

Exclusion Criteria:

* Suffering or any history of disabilities, cardiovascular diseases, asthma, metabolic diseases, etc.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 921 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | Baseline, Month 3

SECONDARY OUTCOMES:
Change in obesity-related anthropometric measurements | Baseline, Month 3
Change in serum lipids and fasting glucose | Baseline，Month 3
Change in dietary and physical activity behaviors | Baseline, Month 3
Change in physical fitness | Baseline, Month 3
Change in percentage of overweight&obesity | Baseline, 3 Month

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Jun Wang, PhD, Study Director — Institute of Child and Adolescent Health,Peking University

REFERENCES:
- [Derived] Li XH, Lin S, Guo H, Huang Y, Wu L, Zhang Z, Ma J, Wang HJ. Effectiveness of a school-based physical activity intervention on obesity in school children: a nonrandomized controlled trial. BMC Public Health. 2014 Dec 16;14:1282. doi: 10.1186/1471-2458-14-1282. PMID 25510313